CLINICAL TRIAL: NCT06328426
Title: Anti-osteoarthritis Therapeutic Potential of Vitamin D With Omega-3 or Metformin: a Randomized Controlled Clinical Trial
Brief Title: Vitamin D With Omega-3 or Metformin in Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Lamiaa Ahmed Abd Elaal Mohammed, Teaching assistant, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Anti-osteoarthritis
Record Dates: First submitted 2024-03-16; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Vitamin D; Docosahexaenoic Acids; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vtamin D and omega-3. (Active Comparator): First arm will be treated with vitamin D and omega-3.
  Interventions: Dietary Supplement: Vitamin D; Dietary Supplement: Omega-3
- vitamin D and metformin (Active Comparator): : Second arm will be treated with vitamin D and metformin.
  Interventions: Dietary Supplement: Vitamin D; Drug: Metformin
- Placebo (Placebo Comparator): Third arm will be treated with placebo.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — The dose of Vitamin D will be 1000 IU /day taken orally. The duration of the intervention will be 4 months.
  Arms: Vtamin D and omega-3.; vitamin D and metformin
Dietary Supplement: Omega-3 — The dose of omega-3 will be 1000 mg /day taken orally. The duration of the intervention will be 4 months.
  Arms: Vtamin D and omega-3.
Drug: Metformin — The dose of metformin will be 1000 IU /day taken orally. The duration of the intervention will be 4 months.
  Arms: vitamin D and metformin
Dietary Supplement: Placebo — The duration of the intervention will be 4 months.
  Arms: Placebo

SUMMARY:
To determine the efficacy of vitamin D with omega-3 or metformin for reducing knee symptoms and effusion synovitis in patients with symptomatic knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA), one of the most common joint diseases, is characterized by fibrosis, rhagadia, ulcers and attrition of articular cartilage due to a number of factors. The aetiology of OA remains unclear, but its occurrence has been associated with age, obesity, inflammation, trauma and genetic factors. The inflammation in OA is distinct from that in rheumatoid arthritis and other autoimmune diseases: it is chronic, comparatively low-grade inflammation, and mediated primarily by the innate immune system. Several studies showed that inflammation triggered by factors like biomechanical stress is involved in the development of osteoarthritis. This stimulates the release of early-stage inflammatory cytokines like interleukin-1 beta (IL-1β), which in turn induces the activation of signaling pathways, such as nuclear factor kappa-light-chain-enhancer of activated B cells (NF-κB), phosphoinositide 3-kinase/protein kinase B. Recently, it has been observed that metabolic syndrome, which is characterized by low-grade inflammation, can increases osteoarthritis risk. Inflammatory cytokines are crucial for the occurrence and progression of OA. The intra-articular proinflammatory and anti-inflammatory cytokines jointly maintain a dynamic balance, in accordance with the physiological metabolism of articular cartilage.

The recent findings highlighting how communication between chondrocytes and macrophages via Damage-associated molecular patterns can maintain the low-grade inflammation (LGI)in the joint microenvironment and initiate the OA process. However, dynamic imbalance between proinflammatory and anti-inflammatory cytokines can cause abnormal metabolism in knee articular cartilage, which leads to deformation, loss and abnormal regeneration, and ultimately destroys the normal structure of the knee joint. The ability of articular cartilage to self-repair once damaged is limited, due to its inability to obtain nutrients from blood vessels, nerves and lymphatic vessels, as well as limitations in the extracellular matrix. Therefore, it has been suggested that the ingredients can inhibit inflammation by reducing the expression and release of inflammatory cytokines(IL-1β , TNF-α, IL -6, IL -15, IL -17 and IL -18 )and enhancing the expression of anti-inflammatory cytokines (IL-4, IGF, IL-10, TGF-β and IL 1RA) which play a cartilage protective role at the gene and protein levels. It holds promise for the development of new disease-modifying therapies for OA.

Current treatments for osteoarthritis only control symptoms and none have been approved by the Food and Drug Administration to prevent or slow the progression of the disease. However, some agents such as vitamin D, Omega 3 and metformin that increase anti-inflammatory cytokines and decrease inflammatory cytokines in OA hold promise for the development of novel disease-modifying therapies.

Vitamin D. Vitamin D seems to reduce chronic inflammation, pathophysiological involved in endothelial dysfunction, its anti-inflammatory actions include downregulation of NF-kB and STAT1/5-mediated signaling, with subsequent down-regulation of the production of anti-inflammatory cytokines, such as TNF-α, IL-1, IL-2β, etc. Moreover, binding of vitamin D to VDR results in the decrease of prostaglandin and cyclooxygenase 2 production, reduction of metalloproteinase-9 (MMP-9) and increase in anti-inflammatory IL-10 production. In animal studies, oral administration of vitamin D significantly reduced OA pain, inflammation, cartilage destruction, and MMPs levels. And in IL-1β stimulated rat chondrocytes revealed that VITD (50, 100, and 500 IU) significantly reduced the mRNA levels of MMPs, NF-κB, TNF-α, and IL-6. Vitamin D was It also was observed that vitamin D attenuated pain and cartilage destruction in OA Animals via enhancing autophagic flux and attenuating Inflammatory Cell Death. Although a conclusive result has not been reached, several randomized control trials indicated that vitamin D supplementation was possible to alleviate pain and improve joint function in knee. Many clinical studies observed that vitamin D2 supplementation can to not only decrease serum levels of LC3A (serum levels of autophagosome protein), inflammatory markers, as well as oxidative stress, but also improve muscle strength and physical performance in patients with knee OA. Other randomized controlled trials have shown that vitamin D supplementation improves oxidative and inflammatory biomarkers, such as total antioxidant capacity, C-reactive protein, and glutathione, but has no effect to others like malondialdehyde and carbonyl group levels.

Omega 3 There is strong evidence that a diet rich in ω-3 fatty acid downregulates markers related to oxidative stress, cartilage degradation, and inflammation in chondrocytes while these markers are elevated with a higher ω-6 fatty acids. Therefore, the quality of polyunsaturated fatty acids (PUFA) might have a distinct role in bone metabolism since metabolites derived from ω-6 and ω-3 fatty acids can act on precursor cells of osteoblast and adipocytes differentially. Some studies suggest that omega-3 fatty acids may have a protective effect on joint cartilage. Cartilage degradation is a key feature of osteoarthritis, and omega-3s may help maintain cartilage integrity by influencing the expression of certain genes and promoting the production of molecules involved in cartilage maintenance. Omega-3 polyunsaturated fatty acids (PUFAs) have been postulated as a potential therapeutic treatment option for individuals with OA. Omega-3 PUFAs are recognized for their anti-inflammatory properties, which could be beneficial in the context of OA to moderate pro-inflammatory markers and cartilage loss.

Metformin In recent years, there has been growing interest in exploring the potential benefits of metformin beyond its use, including its effects on various metabolic and inflammatory conditions, such as osteoarthritis (OA). Considering the existence of metabolic syndrome systemic low-grade inflammation in type knee OA, which accompanying aging, obesity and diabetes, metformin could be considered as a useful and safe component of the personalized therapeutic approach in knee OA patients. In animal studies, metformin has been shown to have ability to the protect cartilage and subchondral bone from damage in mice with collagenase-induced OA (CIOA). In addition, treatment with metformin lowered the level of cartilage biomarkers (CTX-II and COMP). Other studies have suggested that metformin may have protective effects on articular cartilage through the regulation of chondrocyte function and the prevention of cartilage degradation. Metformin activates AMP-activated protein kinase (AMPK), a cellular energy sensor. AMPK activation has been implicated in various cellular processes, including inflammation and cartilage homeostasis. Some researchers suggest that metformin's effects on AMPK activation may contribute to its potential benefits in osteoarthritis. In a cohort study of individuals with diabetes, metformin treatment was associated with a significant reduction in the risk of developing OA).

ELIGIBILITY:
Inclusion Criteria:

2. Are willing to comply with all study related procedures and assessments. 3. Are ambulatory as defined by ability to complete functional performance testing.

4. Radiographic evidence of Kellgren-Lawrence grade II-IV osteoarthritis in one or both knees.

5. Scores 4-10 on the Numerical Rating Scale (NRS) for pain. 6. Stable dose of screening/baseline medications for at least 2 months prior to the anticipated date of study drug dosing.

Exclusion Criteria:

1. Females who are nursing, pregnant or planning to become pregnant during the duration of study drug dosing.
2. Subjects who do not have the capacity to consent themselves.
3. Subjects who are unable to tolerate oral medication.
4. Subjects having previously undergone any of the following treatments in the stated time window:

   1. Surgery on the Study Knee in the past 6 months.
   2. Partial or complete joint replacement in the study knee. Partial or complete joint replacement in the contralateral knee is acceptable if the surgery was performed at least 6 months prior to enrollment and the operative knee is asymptomatic.
   3. Patients who have undergone arthroscopic surgery (including microfracture and meniscectomy) on the Study Knee in the last 2 years prior to the Screening visit or are anticipated to have arthroscopic surgery on either knee at any time during the study period.
   4. Steroid injection, including extended-release corticosteroid (e.g., Zilretta) within the last 5 months.
   5. Biologic (platelet-rich plasma, bone marrow, adipose tissue/cells) or hyaluronic acid injection into the Study Knee in the past 6 months.
5. Subjects with any of the following drug/medication statuses:

   1. Currently taking Losartan.
   2. Currently taking Warfarin or related anticoagulant.
   3. Opioid analgesics taken in the past 8 weeks and are not willing to discontinue these medications through the duration of the study.
   4. Drugs that induce significant cellular stress and are not willing to discontinue these medications through the duration of the study, including alkylating agents, anthracyclines, platins, other chemotherapy drugs.
6. Subjects with any of the following disease statuses:

   1. Significant liver disease (i.e. greater than or equal to 2x the upper limit of normal bilirubin levels).
   2. Significant renal disease (eGFR of <60 ml/min/1.73m2) .
   3. History of other formally diagnosed joint diseases including osteonecrosis, acromegaly, Paget's disease, Ehlers-Danlos Syndrome, Gaucher's disease, Cushing's syndrome, Stickler's syndrome, joint infection, hemophilia, hemochromatosis, or neuropathic arthropathy of any cause.
   4. Any active systemic autoimmune disease with musculoskeletal involvement or any history of system inflammatory arthritis.
   5. Patients with type 1 or 2 diabetes (HbA1c>6.5%) and/or taking medications that affect insulin levels, including: Metformin (within the last week), Glucocorticoids (within the last month), Acarbose (within the last week).
7. Subjects unable to safely practically undergo an MRI (BMI > 40 kg/m2) or size exceeding limits of MRI equipment, implanted metal in study knee near joint surface, incompatible implant/device, severe claustrophobia.
8. Subjects that have any medical condition, including laboratory findings and findings in the medical history or in the pre-study assessments that constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct or evaluation or prevent the patient from fully participating in all aspects of the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Effusion-synovitis volume on musculoskeletal ultrasound. | The measurement will be assessed one day before the treatment and one day after the stoppage of the treatment.
  Ultrasound can reveal Joint space narrowing, subchondral sclerosis, and osteophytosis and changes after intervention.

IPD SHARING:
Plan to Share IPD: Yes
Data will become available to interested investigators upon submitting a reasonable research request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: July, 2026
Access Criteria: Data will become available to interested investigators upon submitting a reasonable research request.